CLINICAL TRIAL: NCT07342582
Title: Identifying the Burden of Hospitalization Due to Rhinovirus (RV) in Children and Mechanisms of Pathogenesis Using Airway Molecular Profiling
Brief Title: The Rhinovirus Hospitalization and Investigation of Nasal-airway Omics (RHINO) Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2025-1076; Protocol Version 12/21/25 (Other: UW Madison); SMPH\PEDIATRICS\INFECT DIS (Other: UW Madison); 1R01AI182200-01A1 (NIH)
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rhinovirus
Keywords: infants; children; symptomatic; asymptomatic; lower respiratory tract infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — liquid media from nasal swabs only, induced sputum, blood, and residual clinical samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Younger Community Cohort (12-36 months of age): Quarterly Surveillance Nasal Swabs and Nasal Swabs targeted around respiratory symptoms for up to 36 months of age, participants will provide one anterior and one mid-turbinate nasal swab sample
  Interventions: Diagnostic Test: Nasal Swab Healthy Surveillance; Diagnostic Test: Nasal Swab Sick Samples; Other: Sick Follow-up Survey
- Hospitalized Cohort of Infants and Children: Generally healthy infants and children hospitalized for respiratory illness will provide one anterior and one mid-turbinate nasal swab sample
  Interventions: Diagnostic Test: Nasal Swab Hospitalized Cohort
- Older Community Cohort (5 to 17 years of age): Age-matched controls for older children in the Hospitalized Group, will be called upon as needed based on enrollment of hospitalized patients
  Interventions: Other: Older Cohort Control Group

INTERVENTIONS:
Diagnostic Test: Nasal Swab Healthy Surveillance — Families will be asked to collect nasal swabs from their children during specified surveillance months (February, April, September, and December). Caregivers will be instructed to only collect surveillance samples during these months if and when children have been free of respiratory symptoms for at least two weeks prior to sampling. Caregiver surveys are part of quarterly surveillance.
  Groups: Younger Community Cohort (12-36 months of age)
Diagnostic Test: Nasal Swab Sick Samples — Caregivers will be instructed to watch for respiratory symptoms and collect nasal swabs 24-48 hours after symptom onset. Caregiver surveys are part of sick sample collection
  Groups: Younger Community Cohort (12-36 months of age)
Diagnostic Test: Nasal Swab Hospitalized Cohort — 2 nasal swabs collected upon consent, one anterior and one mid-turbinate
  Groups: Hospitalized Cohort of Infants and Children
Other: Sick Follow-up Survey — Caregivers are surveyed 7-13 days after sick sample collection
  Groups: Younger Community Cohort (12-36 months of age)
Other: Older Cohort Control Group — Participants will be enrolled as needed based on enrollment of hospitalized patients
  Groups: Older Community Cohort (5 to 17 years of age)

SUMMARY:
The goal of this study is to determine the burden of Rhinoviruses (RVs) as a cause of acute, severe, respiratory illnesses leading to hospitalization. A community cohort of 120 children between 12 and 36 months of age will be enrolled in the first year of the study and followed (when well and sick) for 36 months to identify the circulating RVs and provide samples to establish a host nasal transcriptome differentiating clinical from subclinical RV infections. A hospitalized cohort of 450 infants and children will be enrolled during years 1 through 3 of the study and followed for the duration of their hospitalization to investigate the findings of the community cohort. An additional 100 healthy children aged 5-17 years will be enrolled for age-match comparison with the older hospitalized cohort.

DETAILED DESCRIPTION:
Aim 1: Involves the prospective creation of a cohort of generally healthy children 12 to 36 months to be followed longitudinally for 36 months in an observational study. To determine the frequency of virus infection with RV and other respiratory viruses, children will have two swabs of the nasal mucosa performed whenever they develop an acute respiratory illness (upper respiratory symptoms lasting more than 24 hours) and four times a year for surveillance. One swab will be of the anterior nose and will be used for identification of viruses, and a second mid-turbinate swab will be used for host transcriptomics. This will allow the investigators to create many samples from both symptomatic and asymptomatic infections. The samples will be used to develop a host signature to discriminate symptomatic and asymptomatic infection.

Aim 2a: Involves the evaluation of generally healthy children hospitalized at AFCH with acute, lower respiratory tract infections including bronchiolitis, asthma and community acquired pneumonia. There will also be the evaluation of infants less than 6 months of age who may become ill with an RV syndrome. These children will be evaluated with two nasal swabs as above. This allows the identification of children infected with RV and other respiratory viruses. Application of the host signature developed in Aim 1 will determine the actual proportion of those children who are infected with RV whose illness (clinical symptoms) is caused by RV.

Aim 2b: Involves the prospective creation of a cohort of generally healthy children 5 to 17 years old to be sampled on an as-needed basis to serve as age- and season-matched controls for the Hospitalized Group. To determine the frequency of virus infection with RV and other respiratory viruses, 2 healthy children will provide a single swab of the nasal mucosa within 2 weeks of each hospitalized participant who is 5-17 years of age. The one swab will be of the anterior nose and will be used for identification of viruses. Age matching will occur within 3 groups:

* Ages 5-8 years old: n=50
* Ages 9-13 years old: n=30
* Ages 14-17 years old: n=20

Aim 3: Use parallel bulk and single cell RNA sequencing (scRNA-seq) to identify targetable processes of acute, severe LRT caused by RV. The investigators hypothesize that integrated bulk RNA-sequencing and scRNA-seq will identify immune/inflammatory defects and targets for intervention. Bulk and scRNA-seq on respiratory samples from well-characterized patients with severe RV disease will be performed to test this hypothesis and to compare samples obtained from those with non-severe disease.

ELIGIBILITY:
Inclusion Criteria (Aim 1 and Aim 2b Community Groups):

* Parent/legal guardian is willing and able to provide informed consent in English.
* Willing to comply with all study procedures and be available for the duration of the study.
* Younger Community Group: Generally healthy children 12 to 36 months of age at the time of enrollment
* Older Community Group: Generally healthy children 5 to 17 years of age at the time of enrollment.
* Current patient within primary care system at UW Health

Inclusion Criteria (Aim 2a: Hospitalized Group):

* Parent/legal guardian is willing and able to provide informed consent in English.
* Admitted to American Family Children's Hospital (AFCH) within the past 24 hours
* Children under 18 years of age at the time of enrollment
* Has a diagnosis of bronchiolitis, asthma exacerbation or CAP OR is an infant less than 6 months of age with fever greater than 38 degrees Celsius within 24 hours of hospital admission

Exclusion Criteria (all participants):

* Congenital or currently acquired immunosuppressive condition or medications (e.g., congenital immunodeficiency, Leukemia, Lupus)
* Congenital anomalies that might alter frequency of infection (e.g., unrepaired cleft palate, bronchial cyst, pulmonary sequestration)
* Presence of tracheostomy or gastrostomy tube
* Previously enrolled a different group in the study
* Other child in the same household already enrolled in the study
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Exclusion Criteria (Aim 1: Community Group Only):

* History of chronic pulmonary diseases (e.g., asthma, cystic fibrosis, bronchopulmonary dysplasia (BPD)) (Note: asthma IS exclusionary)
* Acute upper respiratory symptoms within the past week (7 days) at the time of enrollment

Exclusion Criteria (Aim 2: Hospitalized Group Only):

* History of chronic pulmonary diseases, excluding asthma (e.g., cystic fibrosis, bronchopulmonary dysplasia (BPD)) (Note: asthma is NOT exclusionary)
* A positive test for any virus other than RV within the 48 hours prior to and including admission.

Exclusion Criteria (less than 5 years old only (All participants in Aim 1 and some participants in Aim 2a):

* Born prematurely, less than 32 weeks 0 days gestational age

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Aim 1: Generally healthy male and female children 12 to 36 months of age living in Dane County and surrounding areas representative of the general demographics of the county.
  Aim 2a: Hospitalized male and female children between newborn and 17 years of age with acute onset lower respiratory tract infections. These children will span all demographic and socioeconomic groups.
  Aim 2b: Generally healthy male and female children 5 to 17 years of age living in Dane County and surrounding areas representative of the general demographics of the county.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Summary of Rhinovirus Types Identified in Community Cohort | data collected up to 36 months
  To test study hypotheses, the study team will identify the circulating RV types in symptomatic and asymptomatic children.
Aim 1: Unique Nasal Transcriptomic Signature of Clinical Rhinovirus Infections | data collected up to 36 months

SECONDARY OUTCOMES:
Aim 2: Summary of Rhinovirus Types Identified in lower respiratory tract (LRT) infections and upper respiratory tract infections (URI), Reported as Percent in Common | data collected up to 36 months
  To test the hypothesis that there will be an 80 percent overlap between RV types causing acute LRT and URI, investigators will compare all RV types identified in age-matched hospitalized and ambulatory children.
Aim 2: Proportion of Hospitalized Cohort with lower respiratory infections attributable to Rhinovirus | data collected up to 36 months
  The investigators will use host nasal transcriptomics derived from symptomatic and asymptomatic children with RV infection to determine the proportion of age-matched hospitalized LRT infections actually attributable to RV.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the raw RNA-sequencing data will be available in FASTQ files and all of the processed gene counts data and relevant metadata will be available in CSV files. It is customary and expected that the results of this investigation will be published in a scientific journal. All of the data underlying publications will be shared. All raw FASTQ data and aligned counts data will be deposited into the public repository Gene Expression Omnibus (GEO) at the end of the study, so that other researchers can freely make use of the data. The shared data sets will be available in GEO and we will adhere to their guidelines for what the datasets will include.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint by contacting the study team at UW-Madison.